CLINICAL TRIAL: NCT02626182
Title: Evaluation and Treatment of Pulmonary Vascular Disease in Moderate to Severe Cystic Fibrosis Lung Disease
Brief Title: Evaluation and Treatment of Pulmonary Vascular Disease in Moderate to Severe CF
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Jewish Health (Other)
Responsible Party: Principal Investigator, Jennifer Taylor-Cousar, Associate Professor, National Jewish Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NationalJewishHealth
Record Dates: First submitted 2015-12-03; First posted 2015-12-10 (Estimated); Results first posted 2019-07-15 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sildenafil (Experimental): Subjects will be randomized in a 3:1 (sildenafil:placebo) fashion. Subjects randomized to the treatment arm will receive sildenafil 20 mg p.o. t.i.d for 1 week followed by 40 mg p.o. t.i.d. for 11 weeks.
  Interventions: Drug: sildenafil
- Placebo (Placebo Comparator): Subjects randomized to the placebo arm will receive placebo p.o. t.i.d for 1 week followed by 2 placebo tablets p.o. t.i.d. for 11 weeks.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: sildenafil — active sildenafil
  Other Names: Revatio, Viagra
  Arms: Sildenafil
Drug: placebo — sugar pill that looks like sildenafil tablets
  Arms: Placebo

SUMMARY:
This study evaluates the ability of the drug sildenafil to improved exercise capacity, cardiac performance during exercise, and quality of life in patients with moderate to severe CF lung disease. 3/4 of the subjects will receive sildenafil and 1/4 will receive placebo.

DETAILED DESCRIPTION:
Over time, patients with Cystic Fibrosis (CF) develop disabling lung disease that progresses to chronic respiratory failure, exercise intolerance with marked limitation of physical activity, and premature death. Despite substantial improvements in care, patients with CF often develop pulmonary vascular disease (PVD) that leads to pulmonary hypertension. Previous studies have clearly linked severe pulmonary hypertension and right heart failure with high mortality in CF. Early clinical manifestations of PVD prior to the development of cor pulmonale include shortness of breath and dyspnea with exertion, but the extent to which PVD contributes to the decline in exercise tolerance and quality of life in patients with CF is not known. Early evidence of PVD could be recognized in CF patients through standardized exercise testing and echocardiographic evaluation. Identifying those CF patients with PVD prior to the onset of right ventricular dysfunction may allow pharmacologic intervention to attenuate the progression of cardiovascular disease and improve quality of life. Clinical trials have demonstrated that treatment with the phosphodiesterase type 5 inhibitor, sildenafil, can decrease pulmonary vascular resistance and improve exercise tolerance in non-CF patients with pulmonary hypertension. Because experimental and clinical studies have implicated impaired NO-cGMP signaling in the pathophysiology of lung disease in CF, sildenafil may provide a novel pharmacological approach for treating PVD in patients with CF lung disease.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of CF based on the following criteria: Positive sweat chloride ≥60mEq/liter (by pilocarpine iontophoresis) and/or Genotype with two identifiable mutations consistent with CF, and accompanied by one or more clinical features consistent with the CF phenotype
2. Male or female patients ≥ 18 years of age
3. FEV1 ≥ 20% predicted and ≤ 70% predicted (Hankinson)
4. Clinically stable without evidence of acute upper or lower respiratory tract infection or current pulmonary exacerbation within the 14 days prior to the screening visit
5. Ability to reproducibly perform spirometry (according to ATS criteria)
6. Ability to understand and sign a written informed consent or assent and comply with the requirements of the study
7. Willingness to maintain chronic CF medication schedule (e.g. alternating month inhaled antibiotics)

Exclusion Criteria:

1. History of hypersensitivity to sildenafil
2. Use of an investigational agent within the 4-week period prior to Visit 1 (Day 0)
3. Breastfeeding, pregnant, or verbal expression of unwillingness to practice an acceptable birth control method (abstinence, hormonal or barrier methods, partner sterilization or intrauterine device) during participation in the study for women of child-bearing potential.
4. History of significant hepatic disease (AST or ALT > 5 times the upper limit of normal at screening, documented biliary cirrhosis, or portal hypertension),
5. History of significant cardiovascular disease (history of aortic stenosis, coronary artery disease, or life-threatening arrhythmia),
6. History of severe neurological disease (e.g. history of stroke),
7. History of severe hematologic disease (e.g. history of bleeding diathesis; current INR > 2.0
8. History of severe ophthalmologic disease (e.g. history of retinal impairment or non-arteritic ischemic optic neuritis)
9. History of severe renal impairment (creatinine >1.8 mg/dL.)
10. Inability to swallow pills
11. Previous organ transplantation
12. Use of concomitant nitrates, α-blocker, or Ca channel blocker (currently or within one month of Visit 1)
13. Use of concomitant medications known to be potent inhibitors of CYP3A4 [e.g. ketoconazole, itraconazole, ritonavir, clarithromycin, erythromycin, rifampin (currently or within one month of initiation of study drug)] NOTE: use of azithromycin is NOT a cause for exclusion
14. History of sputum or throat swab culture yielding Burkholderia cepacia or Mycobacterium massiliense within 2 years of screening
15. Weight less than 40 kg at Screening
16. History of migraine headaches.
17. Resting room air oxygen saturation <80% without supplemental oxygen
18. Presence of a condition or abnormality that in the opinion of the investigator would compromise the safety of the subject or the quality of the data
19. Start of CFTR modulator therapy less than 1 month prior to first dose of sildenafil or placebo
20. Use of anticoagulants
21. Frank pulmonary hypertension (RVSP >40 mmHg by ECHO)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2015-12; Primary Completion 2018-01-18 (Actual); Study Completion 2018-01-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer L Taylor-Cousar, MD, Principal Investigator — National Jewish Health
Locations (1):
- National Jewish Health, Denver, Colorado, United States

REFERENCES:
- [Background] Orenstein DM, Higgins LW. Update on the role of exercise in cystic fibrosis. Curr Opin Pulm Med. 2005 Nov;11(6):519-23. doi: 10.1097/01.mcp.0000181476.92810.07. PMID 16217178
- [Background] Pianosi P, Leblanc J, Almudevar A. Peak oxygen uptake and mortality in children with cystic fibrosis. Thorax. 2005 Jan;60(1):50-4. doi: 10.1136/thx.2003.008102. PMID 15618583
- [Background] Almajed A, Lands LC. The evolution of exercise capacity and its limiting factors in cystic fibrosis. Paediatr Respir Rev. 2012 Dec;13(4):195-9. doi: 10.1016/j.prrv.2012.01.001. Epub 2012 Feb 10. PMID 23069115
- [Background] Jiang K, Jiao S, Vitko M, Darrah R, Flask CA, Hodges CA, Yu X. The impact of Cystic Fibrosis Transmembrane Regulator Disruption on cardiac function and stress response. J Cyst Fibros. 2016 Jan;15(1):34-42. doi: 10.1016/j.jcf.2015.06.003. Epub 2015 Jun 25. PMID 26119592
- [Background] Galie N, Ghofrani HA, Torbicki A, Barst RJ, Rubin LJ, Badesch D, Fleming T, Parpia T, Burgess G, Branzi A, Grimminger F, Kurzyna M, Simonneau G; Sildenafil Use in Pulmonary Arterial Hypertension (SUPER) Study Group. Sildenafil citrate therapy for pulmonary arterial hypertension. N Engl J Med. 2005 Nov 17;353(20):2148-57. doi: 10.1056/NEJMoa050010. PMID 16291984
- [Background] Mourani PM, Sontag MK, Ivy DD, Abman SH. Effects of long-term sildenafil treatment for pulmonary hypertension in infants with chronic lung disease. J Pediatr. 2009 Mar;154(3):379-84, 384.e1-2. doi: 10.1016/j.jpeds.2008.09.021. Epub 2008 Oct 31. PMID 18950791
- [Background] Montgomery GS, Sagel SD, Taylor AL, Abman SH. Effects of sildenafil on pulmonary hypertension and exercise tolerance in severe cystic fibrosis-related lung disease. Pediatr Pulmonol. 2006 Apr;41(4):383-5. doi: 10.1002/ppul.20393. PMID 16479610
- [Background] Lubamba B, Lecourt H, Lebacq J, Lebecque P, De Jonge H, Wallemacq P, Leal T. Preclinical evidence that sildenafil and vardenafil activate chloride transport in cystic fibrosis. Am J Respir Crit Care Med. 2008 Mar 1;177(5):506-15. doi: 10.1164/rccm.200703-344OC. Epub 2007 Nov 15. PMID 18006891
- [Background] Taylor-Cousar JL, Wiley C, Felton LA, St Clair C, Jones M, Curran-Everett D, Poch K, Nichols DP, Solomon GM, Saavedra MT, Accurso FJ, Nick JA. Pharmacokinetics and tolerability of oral sildenafil in adults with cystic fibrosis lung disease. J Cyst Fibros. 2015 Mar;14(2):228-36. doi: 10.1016/j.jcf.2014.10.006. Epub 2014 Nov 13. PMID 25466700

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sildenafil | Placebo
Started | 11 | 3
Completed | 9 | 3
Not Completed | 2 | 0
Not completed — Adverse Event | 2 | 0

BASELINE CHARACTERISTICS:
Population: All patients who completed all 12 weeks of study drug or placebo are included in the baseline analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sildenafil | Placebo | Total
Number analyzed (Participants) | 9 | 3 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.5 (10.6) | 31.3 (1.5) | 32.2 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 5 | 1 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 9 | 3 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 3 | 0

OUTCOME MEASURES:

1. Primary Outcome: 6 Minute Walk Distance
Description: Change in distance walked between week 1 and week 13 were compared. The difference between the two time points is reported.
Time Frame: Weeks 1, 13
Population: All subjects who received 12 weeks of sildenafil 40 mg po tid or placebo po tid with the exception of 1 extreme outlier in the placebo group who was excluded.
Measure: Mean (Standard Deviation); unit: meters
Groups:
- Sildenafil: Subjects who received sildenafil 40 mg po tid
- Placebo: Subjects who received placebo for 12 weeks
Arm/Group | Sildenafil | Placebo
Number analyzed (Participants) | 9 | 2
meters | 25.2 (18.8) | 0.75 (5.44)

2. Primary Outcome: Cardiopulmonary Exercise Test Work Rate
Description: Work rate (the amount of energy being expended to cycle) was assessed at weeks 1 and 13. The change in maximum work measured during CPET between weeks 1 and 13 is reported.
Time Frame: Weeks 1 and 13
Population: Patients who received sildenafil 40 mg po tid or placebo po tid for 12 weeks
Measure: Mean (Standard Deviation); unit: watts
Arm/Group | Sildenafil | Placebo
Number analyzed (Participants) | 9 | 3
watts | -0.20 (2.96) | -0.27 (4.15)

3. Secondary Outcome: Cystic Fibrosis Quality of Life-Revised Respiratory Domain Score
Description: The CFQ-R Respiratory domain score (scale 0-100 with higher scores indicating better quality of life) was assessed at weeks 1 and 13. The change in the score between week 1 and week 13 is reported.
Time Frame: Assessed at weeks 1 and 13
Population: Subjects who received sildenafil 40 mg po tid or placebo tid for 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sildenafil | Placebo
Number analyzed (Participants) | 9 | 3
units on a scale | 8.62 (18.23) | -9.23 (3.23)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of signing of consent until 2 weeks after the subject's final clinic visit (approximately 5 months)
Arm/Group | Sildenafil | Placebo
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/3
Serious Adverse Events (participants affected / at risk) | 2/9 | 0/3
Other Adverse Events (participants affected / at risk) | 9/9 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sildenafil (N=9) | Placebo (N=3)
Pulmonary exacerbation (Reproductive system and breast disorders) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sildenafil (N=9) | Placebo (N=3)
Sinus congestion (General disorders) | 6 (6) | 1 (1) — Sinus congestion
Flushing (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) — Facial flushing
Cough/congestion (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3)
Epistaxis (General disorders) | 1 (2) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (7) | 0 (0) — Pain
Fever (General disorders) | 2 (2) | 0 (0)
Stomach discomfort (Gastrointestinal disorders) | 2 (2) | 0 (0) — Heartburn/stomach upset
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) — UTI
Tooth pain (General disorders) | 1 (1) | 0 (0) — pericoronitis
Conjuctivitis (Eye disorders) | 1 (1) | 0 (0) — red eyes
Increased sputum (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Wheeze (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Chest pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Shingles (Infections and infestations) | 1 (1) | 0 (0)
Parasthesia (Nervous system disorders) | 1 (2) | 0 (0) — Numbness/tingling

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-31): https://cdn.clinicaltrials.gov/large-docs/82/NCT02626182/Prot_SAP_000.pdf